CLINICAL TRIAL: NCT02966171
Title: A Phase I, Open-label, Multi-center, Dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of HMPL-453 in Patients With Advanced Solid Malignancies
Brief Title: A Dose Escalation Study to Assess the Safety and Tolerability of HMPL-453 in Patients With Advanced Solid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated on 23AUG2018 for safety reasons.
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-453-00AU1
Record Dates: First submitted 2016-10-27; First posted 2016-11-17 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Solid Tumor
Keywords: Advanced Solid Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HMPL-453 (Experimental): Two strengths of HMPL-453 tablets (25 mg and 100 mg based on the free base) will be used for clinical studies. The drug products are coated tablets, which are packaged in white induction sealed HDPE bottles. HMPL-453 will be administered to patients as oral tablet(s) on a daily basis, untill disease progression, intolerable toxicity, or death. Dose levels are to be potentially tested in this study include 25, 50, 100, 200, 300, 400, and 500 mg/day.
  Interventions: Drug: HMPL-453

INTERVENTIONS:
Drug: HMPL-453 — oral administration

SUMMARY:
This is a first-time-in-human, phase I, open-label, dose-escalation study of HMPL-453 in patients with advanced or metastatic solid malignancies who have failed or are intolerable to standard therapies or for whom no standard therapies exist. There are preliminary two stages in this study: a dose-escalation stage (stage 1) and a dose-expansion stage (stage 2). We will decide whether to conduct stage 2 or not one month after the last patient included in stage 1.

DETAILED DESCRIPTION:
Dose-escalation stage (stage 1): Patients participating in the dose-escalation stage will take a single dose of HMPL-453 on Day 1 and will be followed for one week for safety observations. After one week of observation, if no safety issues occur, patients can continue multiple dosing of HMPL-453 QD and start on the DLT assessment cycles. Each cycle consists of 28-days. Patients are required to draw blood samples for PK and safety analysis at specific time points during the treatment.

The 3+3 design will be employed for the dose escalation and MTD determination. To limit the number of patients being exposed to potentially ineffective doses, one patient will be enrolled and dosed in the initial dose cohort. If there are no DLT or < 2 CTCAE grade 2 toxicities occur in the first treatment cycle, then the study will be escalated to the next dose cohort. Otherwise, the trial will revert to a standard 3+3 design.

Dose-Expansion Stage (Stage 2): This stage is to further evaluate the safety, tolerability, PD profile, and preliminary anti-tumor activity of HMPL-453 at the RP2D in approximately 10 patients with advanced solid tumor. Patients with FGFR dysregulated advanced solid tumors, including but not limited to, advanced gastric cancer, advanced urothelial bladder cancer, or advanced cholangiocarcinoma (patients with cancers of the gallbladder or ampulla of Vater are not eligible) are preferred to be enrolled.

Expansion stage will begin after dose-escalation stage is completed and the MTD/RP2D has been determined. Patients will receive HMPL-453 with 28-day treatment cycles until disease progression, death, intolerable toxicity, no longer benefiting from the study treatment per investigator's discretion, or withdrawal of consent, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* In the dose escalation stage, patients with locally advanced, or metastatic solid tumor who have failed, or intolerable to, standard therapies or for whom no standard therapies exist will be enrolled.
* In the dose expansion stage, patients with locally advanced, or metastatic solid tumor and FGFR dysregulation who have failed or intolerable to standard therapies or no standard therapies exist are to be enrolled.
* In the dose escalation stage: evaluable or measurable disease according to RECIST Version 1.1. In the dose expansion stage: measurable disease according to RECIST Version 1.1.
* Life expectancy of at least 12 weeks.
* ECOG performance status of 0 or 1

Exclusion Criteria:

* Prior or current treatment with any selective FGFR inhibitor.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Incidence of DLTs by the NCI CTCAE v4.03 | Cycle 1 (DLT assessment window, 28 days) of multiple dosing peroid

SECONDARY OUTCOMES:
Incidence of AEs, clinically significant laboratory abnormalities, and electrocardiographic (ECG) changes and vital signs | from first dose to 30 days after last dose of study treatment
maximum plasma concentration (Cmax) | from first dose to day 56 of multiple dosing peroid
time to reach maximum concentration (Tmax) | from first dose to day 56 of multiple dosing peroid
terminal half-life (t1/2) | from first dose to day 56 of multiple dosing peroid
area under the concentration-time curve (AUC0-t) | from first dose to day 56 of multiple dosing peroid
apparent clearance (CL/F) | from first dose to day 56 of multiple dosing peroid
Serum phosphate level increases | from first dose to Day 21 of the last treatment cycle
Objective response rate (ORR) | Every 8 weeks while being treated with HMPL-453 (expected average of 16 weeks)
Duration of response (DoR) | Every 8 weeks while being treated with HMPL-453 (expected average of 16 weeks)
Disease Control Rate (DCR) | Every 8 weeks while being treated with HMPL-453 (expected average of 16 weeks)
Change in tumor size | Every 8 weeks while being treated with HMPL-453 (expected average of 16 weeks)
  Tumor size is defined as the sum of the lengths of the longest diameters of the RECIST 1.1 target lesions (TLs). Percentage change in tumor size will be determined for patients with measurable disease at baseline and is derived at each visit by the percentage change in the sum of the diameters of TLs compared to baseline.
Progression free survival (PFS) | Every 8 weeks while being treated with HMPL-453 (expected average of 16 weeks)

OTHER OUTCOMES:
FGFR genetic alterations status | expected average of 16 weeks
  Dose Escalation stage (optional): to retrospectively determine the FGFR genetic alterations in tumor sections for the patients who have either a complete or partial response as per RECIST 1.1.
FGFR pathway inhibition by pERK | from first dose to Day 15 of the first treatment cycle
  Dose expansion stage (optional): explores the FGFR pathway inhibition in the fresh tumor samples pre- and after the treatment of HMPL-453.

CONTACTS AND LOCATIONS:
Overall Officials: Weiss Yang, Study Director — Hutchison Medipharma Limited
Locations (4):
- Australia (4):
  - St Vincent's Cancer Services, Sydney, New South Wales
  - Chris O'Brien Lifehouse, Sydney, New South Wales
  - Peninsula and Southeast Oncology, Frankston, Victoria
  - Monash Medical Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided